CLINICAL TRIAL: NCT01982630
Title: A Phase Ib, Multicenter, Placebo and Active- Comparator-Controlled, Randomized, Double-Blind, Clinical Trial to Evaluate the Safety and Efficacy of MK-8521 Compared to Placebo and a Diabetes Drug in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of the Safety and Efficacy of MK-8521 Compared to Placebo and a Diabetes Drug in Participants With Type 2 Diabetes Mellitus (MK-8521-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8521-003
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1: MK-8521 64/120 μg/day (Experimental): Type 2 diabetes mellitus (T2DM) participants received once daily subcutaneous MK-8521 starting at 64 μg on Days 1 to 7 and escalated to 120 μg on Days 8 to 14.
  Interventions: Drug: MK-8521
- Part 1: MK-8521 34/72 μg/day (Experimental): T2DM participants received once daily subcutaneous MK-8521 starting at 34 μg on Days 1 to 7 and escalated to 72 μg on Days 8 to 14.
  Interventions: Drug: MK-8521
- Part 1: Liraglutide 0.6/1.2/1.8 mg/day (Active Comparator): T2DM participants received once daily subcutaneous liraglutide starting at 0.6 mg on Day 1 and 2, escalated to 1.2 mg on Days 3 to 7, and escalated to 1.8 mg on Days 8 to 14.
  Interventions: Drug: Liraglutide
- Part 1: Placebo for MK-8521 (Placebo Comparator): T2DM participants received once daily subcutaneous placebo for MK-8521 for 14 days.
  Interventions: Drug: Placebo
- Part 2: MK-8521 64/120/180/240/300 µg/day-T2DM (Experimental): T2DM participants received once daily subcutaneous MK-8521 titrated to 300 µg starting at 64 µg and increasing to 120 µg on Day 8, 180 µg on Day 15, 240 µg on Day 20, and 300 µg on Day 25. The total number of dosing days was 29.
  Interventions: Drug: MK-8521
- Part 2: Liraglutide 0.6/1.2/1.8 mg/day-T2DM (Active Comparator): T2DM participants received once daily subcutaneous liraglutide titrated to 1.8 mg starting at 0.6 mg and increasing to 1.2 mg on Day 8, and 1.8 mg on Day 15. The total number of dosing days was 29.
  Interventions: Drug: Liraglutide
- Part 2: Placebo for MK-8521-T2DM (Placebo Comparator): T2DM participants received once daily subcutaneous placebo for MK-8521 for 29 days.
  Interventions: Drug: Placebo
- Part 2: MK-8521 64/120 µg/day-Non-Diabetic Overweight/Obese (Experimental): Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 titrated to 120 µg starting at 64 µg and increasing to 120 µg on Day 8. The total number of dosing days was 14.
  Interventions: Drug: MK-8521

INTERVENTIONS:
Drug: MK-8521
  Arms: Part 1: MK-8521 34/72 μg/day; Part 1: MK-8521 64/120 μg/day; Part 2: MK-8521 64/120 µg/day-Non-Diabetic Overweight/Obese; Part 2: MK-8521 64/120/180/240/300 µg/day-T2DM
Drug: Liraglutide
  Arms: Part 1: Liraglutide 0.6/1.2/1.8 mg/day; Part 2: Liraglutide 0.6/1.2/1.8 mg/day-T2DM
Drug: Placebo
  Arms: Part 1: Placebo for MK-8521; Part 2: Placebo for MK-8521-T2DM

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of MK-8521 given once daily compared to placebo and another diabetes drug in participants with Type 2 diabetes mellitus (T2DM).

This study was modified by a protocol amendment to a 2-part trial to further test the safety and tolerability of MK-8521 at higher doses and to compare MK-8521 pharmacokinetics between participants with T2DM and healthy participants. An additional cohort of T2DM participants and a cohort of non-diabetic obese participants has been added.

ELIGIBILITY:
Inclusion Criteria:

* Male, or female of non-childbearing potential with Type 2 diabetes mellitus (Parts 1 and 2) or non-diabetic (Part 2)
* Body mass index (BMI) between: ≥27 and ≤40 kg/m^2
* A1C (average blood sugar for the past 2 to 3 months) value ≥7.0 and ≤11.0 % (Part 1) or ≥ 6.5 and ≤11.0 % (Part 2) at the time of screening (T2DM participants)
* A1C value <5.7 at the time of screening (non-diabetic subjects in Part 2 only)
* On a stable dose of metformin (≥1000 mg total daily dose) for at least 12 weeks at the time of screening (T2DM participants)

Exclusion Criteria:

* Mentally or legally incapacitated
* History of clinically significant psychiatric disorder of the last 5 years. Participants with situational depression may be enrolled in the trial at the discretion of the Investigator
* History of Type 1 diabetes mellitus or a history of ketoacidosis
* History of clinically significant gastrointestinal, hematological, hepatic, immunological, renal, respiratory, genitourinary or major neurological abnormalities or diseases
* History of cardiovascular disease or cardiac conduction disorder
* History of cancer (malignancy). Exceptions may include adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix or other malignancies which have been successfully treated ≥10 years prior to the pre-screening visit
* History of proliferative diabetic retinopathy or maculopathy
* Clinically significant diabetic autonomic neuropathy
* QTc interval ≥470 msec (for males) or ≥480 msec (for females)
* Clinical significant electrocardiogram (ECG) abnormality
* Positive for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus (HIV)
* On a weight loss program and is not weight-stable (weight stable is defined history of <5% change in body weight in the last 3 months
* On a weight loss medication or has undergone bariatric surgery
* Major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the pretrial (screening) visit
* Participated in another investigational trial within 4 weeks prior to the pretrial (screening) visit
* History of acute or chronic pancreatitis of any etiology
* Mean value for triplicate semi-recumbent systolic blood pressure >160 mm Hg and/or diastolic blood pressure >90 mm Hg (after at least a 10-minute seated rest) and blood pressure is considered unlikely to be below these limits by Day-1 (Randomization) with initiation or adjustment of antihypertensive medication
* Event of severe hypoglycemia with seizure or loss of consciousness in the past 12 months
* Treated with anti-hyperglycemic agents other than metformin within the last 12 weeks
* Previous exposure to any glucagon-like peptide-1 (GLP-1) receptor agonist (e.g. Byetta™, Victoza™ or investigational agents)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2014-10-03 (Actual); Study Completion 2014-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 parts: Part 1 evaluated MK-8521, placebo, and liraglutide in participants with Type 2 diabetes mellitus (T2DM); Part 2 evaluated MK-8521 at higher doses, liraglutide, and placebo in participants with T2DM and MK-8521 in non-diabetic, obese participants.
Pre-assignment Details: Participant flow, baseline characteristic, and outcome measure data are presented by study treatment sequence. Adverse events are presented by the individual doses contained in the study treatment sequence.
Period: Overall Study
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521 | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM | Part 2: MK-8521 64/120 µg/Day-Non-Diabetic Overweight/Obese
Started | 10 | 8 | 13 | 9 | 19 | 14 | 6 | 8
Treated | 9 | 8 | 11 | 9 | 18 | 14 | 6 | 8
Completed | 7 | 8 | 8 | 8 | 16 | 11 | 5 | 8
Not Completed | 3 | 0 | 5 | 1 | 3 | 3 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 0
Not completed — Did Not Receive Drug-Technical Issues | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants. Baseline characteristic data presented by treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521 | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM | Part 2: MK-8521 64/120 µg/Day-Non-Diabetic Overweight/Obese | Total
Number analyzed (Participants) | 10 | 8 | 13 | 9 | 19 | 14 | 6 | 8 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.1 (8.6) | 55.0 (6.4) | 54.5 (8.8) | 51.3 (9.0) | 54.6 (6.0) | 54.6 (7.9) | 52.8 (6.9) | 37.9 (14.1) | 52.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 6 | 11 | 9 | 2 | 2 | 42
  Male | 5 | 6 | 8 | 3 | 8 | 5 | 4 | 6 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 12 | 8 | 11 | 8 | 4 | 4 | 63
  Not Hispanic or Latino | 2 | 0 | 1 | 0 | 8 | 6 | 2 | 4 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 13
  White | 4 | 8 | 13 | 8 | 17 | 10 | 5 | 8 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) in Part 1
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. AEs are presented by individual dose received by participants during titration in an assigned study treatment sequence.
Time Frame: Up to approximately 42 days
Population: The analysis population included all participants in Part 1 who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: MK-8521 64 μg/Day: Type 2 Diabetes Mellitus (T2DM) participants received once daily subcutaneous MK-8521 64 μg/day on Days 1 to 7 as part of the MK-8521 64/120 μg/day treatment group schedule.
- Part 1: MK-8521 120 μg/Day: T2DM participants received once daily subcutaneous MK-8521 120 μg/day on Days 8 to 14 as part of the MK-8521 64/120 μg/day treatment group schedule.
- Part 1: MK-8521 34 μg/Day: T2DM participants received once daily subcutaneous MK-8521 34 μg/day on Days 1 to 7 as part of the MK-8521 34/72 μg/day treatment group schedule.
- Part 1: MK-8521 72 μg/Day: T2DM participants received once daily subcutaneous MK-8521 72 μg/day on Days 8 to 14 as part of the MK-8521 34/72 μg/day treatment group schedule.
- Part 1: Liraglutide 0.6 mg/Day: T2DM participants received once daily subcutaneous liraglutide 0.6 mg on Day 1 and 2 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
- Part 1: Liraglutide 1.2 mg/Day: T2DM participants received once daily subcutaneous liraglutide 1.2 mg on Days 3 to 7 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
- Part 1: Liraglutide 1.8 mg/Day: T2DM participants received once daily subcutaneous liraglutide 1.8 mg on Days 8 to 14 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
Arm/Group | Part 1: MK-8521 64 μg/Day | Part 1: MK-8521 120 μg/Day | Part 1: MK-8521 34 μg/Day | Part 1: MK-8521 72 μg/Day | Part 1: Liraglutide 0.6 mg/Day | Part 1: Liraglutide 1.2 mg/Day | Part 1: Liraglutide 1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 11 | 11 | 8 | 8
Participants | 5 | 5 | 1 | 4 | 2 | 7 | 2 | 5

2. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs) in Part 2
Description: as for outcome 1
Time Frame: Up to approximately 57 days
Population: The analysis population included all participants in Part 2 who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: MK-8521 64 μg/Day: Type 2 Diabetes Mellitus (T2DM) participants received once daily subcutaneous MK-8521 64 µg/day on Days 1 to 7 as part of the MK-8521 64/120/180/240/300 µg/day treatment group schedule.
- Part 2: MK-8521 120 μg/Day: T2DM participants received once daily subcutaneous MK-8521 120 µg/day on Days 8 to 14 as part of the MK-8521 64/120/180/240/300 µg/day treatment group schedule.
- Part 2: MK-8521 180 μg/Day: T2DM participants received once daily subcutaneous MK-8521 180 µg/day on Days 15 to 19 as part of the MK-8521 64/120/180/240/300 µg/day treatment group schedule.
- Part 2: MK-8521 240 μg/Day: T2DM participants received once daily subcutaneous MK-8521 240 µg/day on Days 20 to 24 as part of the MK-8521 64/120/180/240/300 µg/day treatment group schedule.
- Part 2: MK-8521 300 μg/Day: T2DM participants received once daily subcutaneous MK-8521 300 µg/day on Days 25 to 29 as part of the MK-8521 64/120/180/240/300 µg/day treatment group schedule.
- Part 2: Liraglutide 0.6 mg/Day: T2DM participants received once daily subcutaneous liraglutide 0.6 mg on Days 1 to 7 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
- Part 2: Liraglutide 1.2 mg/Day: T2DM participants received once daily subcutaneous liraglutide 1.2 mg on Days 8 to 14 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
- Part 2: Liraglutide 1.8 mg/Day: T2DM participants received once daily subcutaneous liraglutide 1.8 mg on Days 15 to 29 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
- Part 2: MK-8521 64 µg/Day-Non-Diabetic Overweight/Obese: Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 64 µg/day on Days 1 to 7 as part of the MK-8521 64/120 µg/day treatment group schedule.
- Part 2: MK-8521 120 µg/Day-Non-Diabetic Overweight/Obese: Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 120 µg/day hon Days 8 to 14 as part of the MK-8521 64/120 µg/day treatment group schedule.
Arm/Group | Part 2: MK-8521 64 μg/Day | Part 2: MK-8521 120 μg/Day | Part 2: MK-8521 180 μg/Day | Part 2: MK-8521 240 μg/Day | Part 2: MK-8521 300 μg/Day | Part 2: Liraglutide 0.6 mg/Day | Part 2: Liraglutide 1.2 mg/Day | Part 2: Liraglutide 1.8 mg/Day | Part 2: Placebo for MK-8521-T2DM | Part 2: MK-8521 64 µg/Day-Non-Diabetic Overweight/Obese | Part 2: MK-8521 120 µg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 15 | 14 | 13 | 13 | 6 | 8 | 8
Participants | 8 | 14 | 6 | 13 | 8 | 8 | 8 | 12 | 3 | 2 | 4

3. Primary Outcome: Number of Participants Discontinuing Study Drug Due to Adverse Events (AEs) in Part 1
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. Discontinuations are presented by individual dose received by participants during titration in an assigned study treatment sequence.
Time Frame: Up to approximately 14 days
Population: The analysis population included all participants in Part 1 who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: MK-8521 64 μg/Day | Part 1: MK-8521 120 μg/Day | Part 1: MK-8521 34 μg/Day | Part 1: MK-8521 72 μg/Day | Part 1: Liraglutide 0.6 mg/Day | Part 1: Liraglutide 1.2 mg/Day | Part 1: Liraglutide 1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 11 | 11 | 8 | 8
Participants | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants Discontinuing Study Drug Due to Adverse Events (AEs) in Part 2
Description: as for outcome 3
Time Frame: Up to approximately 29 days
Population: The analysis population included all participants in Part 2 who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Liraglutide 1.8 mg/Day: Participants received once daily subcutaneous liraglutide 1.8 mg on Days 15 to 29 as part of the liraglutide 0.6/1.2/1.8 mg/day treatment group schedule.
Arm/Group | Part 2: MK-8521 64 μg/Day | Part 2: MK-8521 120 μg/Day | Part 2: MK-8521 180 μg/Day | Part 2: MK-8521 240 μg/Day | Part 2: MK-8521 300 μg/Day | Part 2: Liraglutide 0.6 mg/Day | Part 2: Liraglutide 1.2 mg/Day | Part 2: Liraglutide 1.8 mg/Day | Part 2: Placebo for MK-8521-T2DM | Part 2: MK-8521 64 µg/Day-Non-Diabetic Overweight/Obese | Part 2: MK-8521 120 µg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 15 | 14 | 13 | 13 | 6 | 8 | 8
Participants | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0

5. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 7 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Semi-recumbent heart rate was assessed at baseline on Day 1; Day 7 at predose, 2, 4, 6, 8, 12, 13, 14, 15, 16, 22 hours postdose; and prior to dosing on Day 8. Heart rate was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged before conducting the statistical analysis. TWA0-24hr was calculated as the area under the measurement-time curve (AUC) divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 7 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 7 dose
Population: The analysis population included a subset of participants who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment according to the underlying scientific model and had data available for the analysis of the endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 6 | 8 | 6 | 8
Beats per minute | 7.19 [3.48 to 10.89] | 1.17 [-2.21 to 4.55] | 7.42 [3.74 to 11.09] | 5.69 [2.39 to 8.99]
Statistical Analysis 1: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; Fixed effects for treatment, day and treatment by day interaction, a random effect for participant and baseline TWA0-24hr of heart rate as a covariate; Difference of Least Squares Means = -0.23, 90% CI 2-sided [-4.59 to 4.13]
Statistical Analysis 2: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -6.25, 90% CI 2-sided [-10.48 to -2.01]
Statistical Analysis 3: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: MK-8521 34/72 μg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 6.02, 90% CI 2-sided [1.81 to 10.22]
Statistical Analysis 4: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 1.50, 90% CI 2-sided [-2.65 to 5.64]
Statistical Analysis 5: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -4.52, 90% CI 2-sided [-8.52 to -0.52]
Statistical Analysis 6: Comparison: Part 1: Liraglutide 0.6/1.2/1.8 mg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 1.73, 90% CI 2-sided [-2.38 to 5.83]

6. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 7 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 7: predose, 2, 4, 6, 8, 12, and 16 hours postdose; and prior to dosing on Day 8. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 7 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 7 dose
Population: The analysis population included a subset of participants who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment according to the underlying scientific model and had data available for the analysis of the endpoint. Per-protocol, non-diabetic overweight/obese participants were not planned for the TWA0-24hr analysis of heart rate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Groups:
- Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM: Type 2 diabetes mellitus (T2DM) participants received once daily subcutaneous MK-8521 titrated to 300 µg starting at 64 µg and increasing to 120 µg on Day 8, 180 µg on Day 15, 240 µg on Day 20, and 300 µg on Day 25. The total number of dosing days was 29.
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 6
Beats per minute | 1.99 [0.10 to 3.88] | 4.10 [1.87 to 6.34] | -0.54 [-3.80 to 2.73]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -2.11, 90% CI 2-sided [-4.55 to 0.32]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 2.53, 90% CI 2-sided [-0.61 to 5.66]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 4.64, 90% CI 2-sided [1.35 to 7.93]

7. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 14 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 14: predose, 2, 4, 6, 8, 12, 13, 14, 15, 16, 22 hours postdose and prior to dosing on Day 15. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 14 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 14 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 6 | 8 | 6 | 8
Beats per minute | 9.67 [5.97 to 13.37] | 3.90 [0.52 to 7.28] | 10.32 [6.65 to 14.00] | 9.81 [6.51 to 13.12]
Statistical Analysis 1: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -0.65, 90% CI 2-sided [-5.01 to 3.71]
Statistical Analysis 2: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -6.42, 90% CI 2-sided [-10.66 to -2.19]
Statistical Analysis 3: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: MK-8521 34/72 μg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 5.77, 90% CI 2-sided [1.57 to 9.97]
Statistical Analysis 4: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -0.15, 90% CI 2-sided [-4.29 to 4.00]
Statistical Analysis 5: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -5.91, 90% CI 2-sided [-9.91 to -1.92]
Statistical Analysis 6: Comparison: Part 1: Liraglutide 0.6/1.2/1.8 mg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 0.51, 90% CI 2-sided [-3.60 to 4.62]

8. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 14 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 14: predose, 2, 4, 6, 8, 12, 16, hours postdose; and prior to dosing on Day 15. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 14 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 14 dose
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
Beats per minute | 5.05 [2.79 to 7.30] | 5.93 [3.27 to 8.60] | -0.20 [-4.32 to 3.93]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -0.89, 90% CI 2-sided [-3.80 to 2.02]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 5.24, 90% CI 2-sided [1.34 to 9.15]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 6.13, 90% CI 2-sided [2.05 to 10.22]

9. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 19 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 19: predose, 2, 4, 6, 8, 12, 16, hours post dose; and prior to dosing on Day 20. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 19 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 19 dose
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
Beats per minute | 5.62 [3.19 to 8.05] | 6.20 [3.32 to 9.07] | -2.14 [-6.66 to 2.37]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = -0.57, 90% CI 2-sided [-3.71 to 2.57]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 7.77, 90% CI 2-sided [3.50 to 12.03]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 8.34, 90% CI 2-sided [3.89 to 12.79]

10. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 24 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 24: predose, 2, 4, 6, 8, 12, 16, hours postdose; and prior to dosing on Day 25. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 24 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 24 dose
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 17 | 11 | 5
Beats per minute | 7.30 [4.43 to 10.17] | 5.95 [2.50 to 9.41] | -0.99 [-6.28 to 4.29]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 1.35, 90% CI 2-sided [-2.40 to 5.09]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 8.29, 90% CI 2-sided [3.29 to 13.30]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 6.95, 90% CI 2-sided [1.69 to 12.20]

11. Primary Outcome: Change From Baseline in Time-weighted Average From 0 to 24 Hours (TWA0-24hr) of Heart Rate (HR) After 29 Days of Treatment in Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent HR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; and Day 29: predose, 2, 4, 6, 8, 12, 16 and 24 hours postdose. The repeated measurements were averaged before conducting the analysis. TWA0-24hr was calculated as the AUC divided by the time period of over which the measurements were made (i.e. 24 hrs.). Change from baseline TWA0-24hr HR was calculated as the TWA0-24hr HR at Day 29 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 29 dose
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
Beats per minute | 8.30 [5.31 to 11.29] | 5.84 [2.26 to 9.43] | -1.31 [-6.81 to 4.19]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 2.46, 90% CI 2-sided [-1.42 to 6.34]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 9.61, 90% CI 2-sided [4.42 to 14.81]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 5, analysis 1]; Difference of Least Squares Means = 7.15, 90% CI 2-sided [1.70 to 12.60]

12. Primary Outcome: Change From Baseline in Peak Heart Rate (PHR) at Day 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: PHR was defined as the maximum time matched baseline adjusted heart rate over 24 hours. Semi-recumbent PHR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 7: predose, 2, 4, 6, 8, 12, and 16 hours postdose; and prior to dosing on Day 8. The repeated measurements were averaged before conducting the analysis. Change from baseline PHR was calculated as the peak heart rate at Day 7 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 7 dose
Population: The analysis population included a subset of participants who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment according to the underlying scientific model and had data available for the analysis of the endpoint. Per-protocol, non-diabetic overweight/obese participants were not planned for the analysis of peak heart rate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 6
Beats per minute | 7.94 [5.76 to 10.13] | 11.91 [9.30 to 14.53] | 8.65 [4.86 to 12.43]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; Fixed effects for treatment, day and treatment by day interaction, a random effect for participant and baseline peak heart rate as a covariate; Difference of Least Squares Means = -3.97, 90% CI 2-sided [-6.80 to -1.14]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = -0.70, 90% CI 2-sided [-4.33 to 2.93]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 3.26, 90% CI 2-sided [-0.54 to 7.06]

13. Primary Outcome: Change From Baseline in Peak Heart Rate (PHR) at Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: PHR was defined as the maximum time matched baseline adjusted heart rate over 24 hours. Semi-recumbent PHR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 14: predose, 2, 4, 6, 8, 12, and 16 hours postdose; and prior to dosing on Day 15. The repeated measurements were averaged before conducting the analysis. Change from baseline PHR was calculated as the peak heart rate at Day 14 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 14 dose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 6
Beats per minute | 11.41 [8.50 to 14.32] | 13.00 [9.58 to 16.41] | 8.90 [3.87 to 13.93]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = -1.58, 90% CI 2-sided [-5.31 to 2.15]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 2.52, 90% CI 2-sided [-2.32 to 7.35]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 4.10, 90% CI 2-sided [-0.96 to 9.16]

14. Primary Outcome: Change From Baseline in Peak Heart Rate (PHR) at Day 19 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: PHR was defined as the maximum time matched baseline adjusted heart rate over 24 hours. Semi-recumbent PHR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 19: predose, 2, 4, 6, 8, 12, and 16 hours postdose; and prior to dosing on Day 20. The repeated measurements were averaged before conducting the analysis. Change from baseline PHR was calculated as the peak heart rate at Day 19 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 19 dose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
Beats per minute | 11.26 [8.28 to 14.24] | 14.75 [11.25 to 18.25] | 7.30 [2.00 to 12.61]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = -3.48, 90% CI 2-sided [-7.31 to 0.34]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 3.96, 90% CI 2-sided [-1.11 to 9.03]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 7.44, 90% CI 2-sided [2.16 to 12.73]

15. Primary Outcome: Change From Baseline in Peak Heart Rate (PHR) at Day 24 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: PHR was defined as the maximum time matched baseline adjusted heart rate over 24 hours. Semi-recumbent PHR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; Day 24: predose, 2, 4, 6, 8, 12, and 16 hours postdose; and prior to dosing on Day 25. The repeated measurements were averaged before conducting the analysis. Change from baseline PHR was calculated as the peak heart rate at Day 24 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 24 dose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 17 | 11 | 5
Beats per minute | 14.09 [10.60 to 17.57] | 14.06 [9.85 to 18.27] | 9.39 [3.03 to 15.76]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 0.03, 90% CI 2-sided [-4.51 to 4.57]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 4.70, 90% CI 2-sided [-1.33 to 10.73]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 4.66, 90% CI 2-sided [-1.67 to 11.00]

16. Primary Outcome: Change From Baseline in Peak Heart Rate (PHR) at Day 29 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: PHR was defined as the maximum time matched baseline adjusted heart rate over 24 hours. Semi-recumbent PHR was measured in triplicate with at least a 1-2-minute interval between measurements at the following time points: baseline on Day 1; and Day 29: predose 2, 4, 6, 8, 12, 16, and 24 hours post dose. The repeated measurements were averaged before conducting the analysis. Change from baseline PHR was calculated as the peak heart rate at Day 29 minus baseline where baseline was defined as predose on Day 1.
Time Frame: Baseline (predose Day 1) and up to 24 hours post Day 29 dose
Population: as for outcome 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
Beats per minute | 16.01 [12.88 to 19.13] | 12.66 [8.91 to 16.41] | 7.13 [1.49 to 12.76]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 3.34, 90% CI 2-sided [-0.70 to 7.39]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 8.88, 90% CI 2-sided [3.53 to 14.23]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 12, analysis 1]; Difference of Least Squares Means = 5.54, 90% CI 2-sided [-0.08 to 11.15]

17. Primary Outcome: Change From Baseline in Resting Morning Heart Rate (RMHR) After the Day 7 Dose for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent RMHR was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged for each time point. Change from baseline RMHR was calculated as the RMHR 24 hours after the Day 7 dose (predose Day 8) minus baseline. Baseline was an average of 2 readings prior to dosing on Day 1.
Time Frame: Baseline (predose Day 1) and Day 8 (24 hours after Day 7)
Population: The analysis population included a subset of participants who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment according to the underlying scientific model and had data available for the analysis of the endpoint. Per-protocol, non-diabetic overweight/obese participants were not planned for the analysis of resting morning heart rate.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 6
Beats per minute | 1.65 [-1.00 to 4.29] | 5.20 [2.07 to 8.33] | 0.59 [-3.99 to 5.18]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; Fixed effects for treatment, day and treatment by day interaction, a random effect for participant and baseline RMHR as a covariate; Difference of Least Squares Means = -3.55, 90% CI 2-sided [-6.98 to -0.12]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 1.05, 90% CI 2-sided [-3.38 to 5.49]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 4.61, 90% CI 2-sided [-0.02 to 9.23]

18. Primary Outcome: Change From Baseline in Resting Morning Heart Rate (RMHR) After the Day 14 Dose for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent RMHR was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged for each time point. Change from baseline RMHR was calculated as the RMHR 24 hours after the Day 14 dose (predose Day 15) minus baseline. Baseline was an average of 2 readings prior to dosing on Day 1.
Time Frame: Baseline (predose Day 1) and Day 15 (24 hours after Day 14)
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
Beats per minute | 4.22 [1.58 to 6.87] | 5.38 [2.25 to 8.51] | -4.42 [-9.32 to 0.47]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = -1.16, 90% CI 2-sided [-4.59 to 2.28]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 8.65, 90% CI 2-sided [3.99 to 13.31]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 9.80, 90% CI 2-sided [4.96 to 14.65]

19. Primary Outcome: Change From Baseline in Resting Morning Heart Rate (RMHR) After the Day 19 Dose for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent RMHR was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged for each time point. Change from baseline RMHR was calculated as the RMHR 24 hours after the Day 19 dose (predose Day 20) minus baseline. Baseline was an average of 2 readings prior to dosing on Day 1.
Time Frame: Baseline (predose Day 1) and Day 20 (24 hours after Day 19)
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 12 | 5
Beats per minute | 6.41 [3.76 to 9.05] | 10.44 [7.24 to 13.65] | -3.82 [-8.72 to 1.07]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = -4.04, 90% CI 2-sided [-7.52 to -0.56]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 10.23, 90% CI 2-sided [5.57 to 14.89]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 14.27, 90% CI 2-sided [9.38 to 19.15]

20. Primary Outcome: Change From Baseline in Resting Morning Heart Rate (RMHR) After the Day 24 Dose for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent RMHR was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged for each time point. Change from baseline RMHR was calculated as the RMHR 24 hours after the Day 24 dose (predose Day 25) minus baseline. Baseline was an average of 2 readings prior to dosing on Day 1.
Time Frame: Baseline (predose Day 1) and Day 25 (24 hours after Day 24)
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
Beats per minute | 7.51 [4.77 to 10.25] | 9.63 [6.35 to 12.91] | -5.82 [-10.72 to -0.93]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = -2.12, 90% CI 2-sided [-5.70 to 1.47]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 13.34, 90% CI 2-sided [8.64 to 18.03]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 15.45, 90% CI 2-sided [10.53 to 20.38]

21. Primary Outcome: Change From Baseline in Resting Morning Heart Rate (RMHR) After the Day 29 Dose for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: Semi-recumbent RMHR was measured in triplicate with at least a 1-2-minute interval between measurements. The repeated measurements were averaged for each time point. Change from baseline RMHR was calculated as the RMHR 24 hours after the Day 29 dose minus baseline. Baseline was an average of 2 readings prior to dosing on Day 1.
Time Frame: Baseline (predose Day 1) and Day 30 (24 hours after Day 29)
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
Beats per minute | 9.41 [6.67 to 12.15] | 7.30 [4.01 to 10.58] | -1.02 [-5.92 to 3.87]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 2.11, 90% CI 2-sided [-1.47 to 5.70]
Statistical Analysis 2: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 10.43, 90% CI 2-sided [5.73 to 15.13]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 17, analysis 1]; Difference of Least Squares Means = 8.32, 90% CI 2-sided [3.40 to 13.24]

22. Primary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours (AUC0-24hr) of MK-8521 on Days 1, 7, and 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: AUC0-24hr was the area under the concentration-time curve of MK-8521 from time zero to 24 hours after administration. Plasma samples were collected from predose to 24 hours postdose for determination of AUC0-24hr. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. AUC0-24hr is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1, 7, and 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hour
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 9 | 8
nM•hour
  Day 1 | 6.11 (47.6) | 2.25 (27.5)
  Day 7: number analyzed (Participants) | 7 | 8
  Day 7 | 14.4 (55.9) | 5.63 (24.6)
  Day 14: number analyzed (Participants) | 7 | 8
  Day 14 | 32.8 (42.8) | 12.6 (26.6)

23. Primary Outcome: Maximum Concentration (Cmax) of MK-8521 on Days 1 and 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Cmax was the maximum observed concentration of MK-8521 in plasma after administration. Plasma samples were collected from predose to 24 hours postdose for determination of Cmax. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. Cmax is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 9 | 8
nM
  Day 1 | 0.350 (41.4) | 0.128 (21.4)
  Day 7: number analyzed (Participants) | 7 | 8
  Day 7 | 0.710 (57.6) | 0.275 (31.2)

24. Primary Outcome: Maximum Concentration (Cmax) of MK-8521 on Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Cmax was the maximum observed concentration of MK-8521 in plasma after administration on Day 14. Plasma samples were collected from predose to 120 hours postdose for determination of Cmax. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. Cmax is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, 24, 72, 96, and 120 hours post-dose on Day 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
nM | 1.70 (38.4) | 0.619 (27.0)

25. Primary Outcome: Trough Concentration (Ctrough) of MK-8521 on Days 1, 7, and 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Ctrough was the lowest observed concentration of MK-8521 in plasma. Plasma samples were collected predose on Day 2 (sampled after the Day 1 dose and prior to Day 2 dose), 7, and 14 for determination of Ctrough. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. Ctrough is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose on Days 2, 7, and 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 9 | 8
nM
  Day 1 | 0.322 (33.2) | 0.119 (20.6)
  Day 7: number analyzed (Participants) | 7 | 8
  Day 7 | 0.442 (83.6) | 0.207 (21.8)
  Day 14: number analyzed (Participants) | 7 | 8
  Day 14 | 1.16 (43.3) | 0.506 (27.5)

26. Primary Outcome: Time to Maximum Concentration (Tmax) of MK-8521 on Days 1 and 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Tmax was the time required to reach the maximum concentration of MK-8521 in plasma. Plasma samples were collected from predose to 24 hours postdose for determination of Tmax. Tmax is presented as median with a full range.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 9 | 8
Hours
  Day 1 | 16 [10 to 24] | 16 [10 to 24]
  Day 7: number analyzed (Participants) | 7 | 8
  Day 7 | 7 [6 to 10] | 6 [1 to 10]

27. Primary Outcome: Time to Maximum Concentration (Tmax) of MK-8521 on Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Tmax was the time required to reach the maximum concentration of MK-8521 in plasma. Plasma samples were collected from predose to 120 hours postdose for determination of Tmax. Tmax is presented as median with a full range.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, 24, 72, 96, and 120 hours post-dose on Day 14
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
Hours | 8 [1 to 8] | 6 [4 to 12]

28. Primary Outcome: Apparent Terminal Half Life (t1/2) of MK-8521 on Days 1 and 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: t1/2 was the time required to divide the MK-8521 concentration by half after reaching pseudo-equilibrium. Plasma samples were collected from predose to 24 hours postdose for determination of t1/2. t1/2 is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: The analysis population included a subset of participants who complied with the protocol sufficiently to ensure that their data exhibited the effects of treatment according to the underlying scientific model and had data available for the analysis of the endpoint. t1/2 was not measured for Days 1 and 7 since terminal phase was not adequately captured with sampling times up to 24 hours post dose.
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Apparent Terminal Half Life (t1/2) of MK-8521 on Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: t1/2 was the time required to divide the MK-8521 concentration by half after reaching pseudo-equilibrium. Plasma samples were collected from predose to 120 hours postdose for determination of t1/2. t1/2 was measured on Day 14 which is the longest time point for sampling for T2DM participants in Part 1. t1/2 is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, 24, 72, 96, and 120 hours post-dose on Day 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
Hours | 15.6 (16.1) | 17.2 (17.0)

30. Primary Outcome: Accumulation Ratio of the Area Under the Concentration-time Curve From 0 to 24 Hours (AUC0-24hr) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Plasma samples were collected from predose to 24 hours postdose for determination of the accumulation ratio of AUC0-24hr. The geometric mean accumulation ratio was calculated as Day 7 AUC0-24hr/Day 1 AUC0-24hr and presented as geometric mean ratio with a full range.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: as for outcome 5
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
Ratio | 2.31 [1.85 to 2.66] | 2.50 [1.80 to 3.73]

31. Primary Outcome: Accumulation Ratio of the Maximum Concentration (Cmax) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Plasma samples were collected from predose to 24 hours postdose for determination of the accumulation ratio of Cmax. The geometric mean accumulation ratio was calculated as Day 7 Cmax/Day 1 Cmax and presented as geometric mean ratio with a full range.
Time Frame: Predose and 1, 2, 4, 6, 8, 10, 12, 16, and 24 hours post-dose on Days 1 and 7
Population: as for outcome 5
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
Ratio | 2.00 [1.41 to 2.35] | 2.14 [1.61 to 2.83]

32. Primary Outcome: Accumulation Ratio of the Trough Concentration (Ctrough) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: Plasma samples were collected predose on Days 2 (sampled after the Day 1 dose and prior to Day 2 dose) and 7 for determination of the accumulation ratio of Ctrough. The geometric mean accumulation ratio was calculated as Day 7 Ctrough/Day 1 Ctrough (sampled after the Day 1 dose and prior to Day 2 dose) and presented as geometric mean ratio with a full range.
Time Frame: Predose on Days 2 and 7
Population: as for outcome 5
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day
Number analyzed (Participants) | 7 | 8
Ratio | 1.37 [0.39 to 2.13] | 1.73 [1.46 to 1.93]

33. Primary Outcome: Area Under the Concentration-time Curve From 0 to 24 Hours (AUC0-24hr) of MK-8521 on Days 1, 7, and 14 for Type 2 Diabetes Mellitus (T2DM) and Non-Diabetic Overweight/Obese Participants in Part 2
Description: as for outcome 22
Time Frame: Predose and 1, 2, 6, 10, 16, and 24 hours postdose on Days 1, 7, and 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM•hour
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: MK-8521 64/120 µg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 8
nM•hour
  Day 1 | 6.46 (49.5) | 7.68 (34.8)
  Day 7 | 15.1 (35.6) | 15.0 (35.9)
  Day 14 | 30.0 (35.8) | 34.4 (19.5)

34. Primary Outcome: Accumulation Ratio of the Area Under the Concentration-time Curve From 0 to 24 Hours (AUC0-24hr) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) and Non-Diabetic Overweight/Obese Participants in Part 2
Description: Plasma samples were collected from predose to 24 hours postdose for determination of the accumulation ratio of AUC0-24hr. The geometric mean accumulation ratio was calculated as Day 7 AUC0-24hr/Day 1 AUC0-24hr and presented as geometric mean ratio and percent geometric coefficient of variation.
Time Frame: Predose and 1, 2, 6, 10, 16, and 24 hours post-dose on Days 1 and 7
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: MK-8521 64/120 µg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 8
Ratio | 2.33 (22.2) | 1.95 (28.6)

35. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: FPG was measured predose on Days 1 and 7. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 7. FPG is presented as mean change from baseline with a standard error.
Time Frame: Predose on Days 1 (baseline) and 7
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Part 1: Placebo for MK-8521: Participants received once daily subcutaneous placebo for MK-8521 for 14 days.
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 7 | 8 | 9 | 8
mg/dL | -23.57 (10.75) | -39.00 (8.44) | -59.11 (7.09) | -11.13 (7.26)

36. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: FPG was measured predose on Days 1 and 14. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 14. FPG is presented as mean change from baseline with a standard error.
Time Frame: Predose on Days 1 (baseline) and 14
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 7 | 8 | 8 | 8
mg/dL | -41.29 (11.22) | -48.50 (13.21) | -59.25 (4.98) | -13.50 (9.54)

37. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 7 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Blood samples for glucose were collected immediately prior to, and after each meal. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Blood for plasma glucose concentrations was obtained at predose Day 1 at pre meal (breakfast), 0.5, 1, 2, 3, 4 (pre lunch), 4.5, 5, 6, 7, 10 (pre dinner), 10.5, 11, 12, 13, 15 and 23 hours post breakfast meal; and on Day 7 at 1 (pre breakfast), 1.5, 2, 3, 4, 5 (pre lunch), 5.5, 6, 7, 8, 11 (pre dinner), 11.5, 12, 13, 14, 16, 24 hours post dose. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with fixed effects for treatment, day and treatment by day interaction, a random effect for participant, and baseline 24-hour WMG as a covariate. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 7 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 6 | 8 | 6 | 8
mg/dL | -24.08 [-45.46 to -2.71] | -27.54 [-46.39 to -8.69] | -53.64 [-75.20 to -32.08] | 2.36 [-16.20 to 20.92]
Statistical Analysis 1: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; Fixed effects for treatment, day and treatment by day interaction, a random effect for participant and baseline 24-hour WMG as a covariate; Difference of Least Squares Means = 29.56, 90% CI 2-sided [4.34 to 54.77]
Statistical Analysis 2: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 26.10, 90% CI 2-sided [2.02 to 50.19]
Statistical Analysis 3: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: MK-8521 34/72 μg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 3.45, 90% CI 2-sided [-20.23 to 27.14]
Statistical Analysis 4: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -26.45, 90% CI 2-sided [-49.96 to -2.93]
Statistical Analysis 5: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -29.90, 90% CI 2-sided [-52.04 to -7.77]
Statistical Analysis 6: Comparison: Part 1: Liraglutide 0.6/1.2/1.8 mg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -56.00, 90% CI 2-sided [-79.53 to -32.48]

38. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 1
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Blood samples for glucose were collected immediately prior to and after each meal. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Blood for plasma glucose concentrations was obtained on Day -1 at pre meal (breakfast), 0.5, 1, 2, 3, 4 (pre lunch), 4.5, 5, 6, 7, 10 (pre dinner), 10.5, 11, 12, 13, 15 and 23 hours post breakfast meal; and on Day 14 at 1 (pre breakfast), 1.5, 2, 3, 4, 5 (pre lunch), 5.5, 6, 7, 8, 11(pre dinner), 11.5, 12, 13, 14, 16, 24 hours post dose. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with fixed effects for treatment, day and treatment by day interaction, a random effect for participant, and baseline 24-hour WMG as a covariate. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 14 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1: MK-8521 64/120 μg/Day | Part 1: MK-8521 34/72 μg/Day | Part 1: Liraglutide 0.6/1.2/1.8 mg/Day | Part 1: Placebo for MK-8521
Number analyzed (Participants) | 6 | 8 | 6 | 8
mg/dL | -37.24 [-58.61 to -15.86] | -45.63 [-64.49 to -26.78] | -52.20 [-73.76 to -30.64] | -2.00 [-20.56 to 16.56]
Statistical Analysis 1: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 14.96, 90% CI 2-sided [-10.25 to 40.18]
Statistical Analysis 2: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Liraglutide 0.6/1.2/1.8 mg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 6.57, 90% CI 2-sided [-17.52 to 30.65]
Statistical Analysis 3: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: MK-8521 34/72 μg/Day; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 8.40, 90% CI 2-sided [-15.29 to 32.08]
Statistical Analysis 4: Comparison: Part 1: MK-8521 64/120 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -35.23, 90% CI 2-sided [-58.75 to -11.72]
Statistical Analysis 5: Comparison: Part 1: MK-8521 34/72 μg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -43.63, 90% CI 2-sided [-65.77 to -21.50]
Statistical Analysis 6: Comparison: Part 1: Liraglutide 0.6/1.2/1.8 mg/Day vs Part 1: Placebo for MK-8521; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -50.20, 90% CI 2-sided [-73.72 to -26.68]

39. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: FPG was measured predose on Days 1 and 14. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 14. FPG is presented as least squares mean change from baseline with a 95% confidence interval.
Time Frame: Predose on Days 1 (baseline) and 14
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
mg/dL | -45.89 [-56.44 to -35.33] | -39.80 [-48.27 to -31.33] | -14.69 [-43.93 to 14.55]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; Fixed effects for treatment, day and treatment by day interaction, a random effect for participant and baseline FPG as a covariate; Difference of Least Squares Means = -31.20, 90% CI 2-sided [-56.59 to -5.81]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -25.12, 90% CI 2-sided [-50.25 to 0.01]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -6.08, 90% CI 2-sided [-17.31 to 5.14]

40. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 19 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: FPG was measured predose on Days 1 and 19. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 19. FPG is presented as least squares mean change from baseline with a 95% confidence interval.
Time Frame: Predose on Days 1 (baseline) and 19
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
mg/dL | -44.22 [-54.77 to -33.66] | -47.33 [-55.80 to -38.86] | -16.74 [-45.98 to 12.51]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -27.48, 90% CI 2-sided [-52.87 to -2.09]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -30.59, 90% CI 2-sided [-55.72 to -5.46]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = 3.11, 90% CI 2-sided [-8.11 to 14.34]

41. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 24 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: FPG was measured predose on Days 1 and 24. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 24. FPG is presented as least squares mean change from baseline with a 95% confidence interval.
Time Frame: Predose on Days 1 (baseline) and 24
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 17 | 11 | 5
mg/dL | -40.14 [-51.00 to -29.27] | -50.14 [-59.30 to -40.99] | -44.73 [-73.97 to -15.49]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = 4.59, 90% CI 2-sided [-20.88 to 30.06]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -5.42, 90% CI 2-sided [-30.68 to 19.85]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = 10.01, 90% CI 2-sided [-1.77 to 21.78]

42. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 29 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: FPG was measured predose on Days 1 and 29. The change from baseline of FPG was calculated as the difference between the predose measurement on Day 1 (baseline) and the measurement obtained predose on Day 29. FPG is presented as least squares mean change from baseline with a 95% confidence interval.
Time Frame: Predose on Days 1 (baseline) and 29
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
mg/dL | -52.54 [-63.74 to -41.33] | -52.06 [-61.21 to -42.91] | -37.55 [-66.80 to -8.31]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -14.98, 90% CI 2-sided [-40.53 to 10.57]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -14.50, 90% CI 2-sided [-39.77 to 10.76]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 39, analysis 1]; Difference of Least Squares Means = -0.48, 90% CI 2-sided [-12.47 to 11.52]

43. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 14 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Plasma glucose concentrations were obtained on Day -1 at pre meal (breakfast), 1, 3, 4 (pre lunch), 5, 7, 10 (pre dinner), 11, 13, 15 and 23 hours post breakfast meal and Day 14 at 1 (pre breakfast), 2, 4, 5 (pre lunch), 6, 8, 11 (pre dinner), 12, 14, 16, 24 hours post dose. The timing of samples on Day -1 are relative to the breakfast meal. Day 14 samples are relative to dosing. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with group, day and group by day interaction as fixed effects, baseline 24-hour WMG as a covariate, and participant as a random effect. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 14 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
mg/dL | -47.52 [-56.82 to -38.22] | -51.24 [-58.02 to -44.45] | -3.84 [-30.31 to 22.63]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -43.68, 90% CI 2-sided [-65.81 to -21.55]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -47.40, 90% CI 2-sided [-69.35 to -25.45]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 3.72, 90% CI 2-sided [-5.76 to 13.19]

44. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 19 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Plasma glucose concentrations were obtained on Day -1 at pre meal (breakfast), 1, 3, 4 (pre lunch), 5, 7, 10 (pre dinner), 11, 13, 15 and 23 hours post breakfast meal and Day 19 at 1 (pre breakfast), 2, 4, 5 (pre lunch), 6, 8, 11 (pre dinner), 12, 14, 16, 24 hours post dose. The timing of samples on Day -1 are relative to the breakfast meal. Day 19 samples are relative to dosing. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with group, day and group by day interaction as fixed effects, baseline 24-hour WMG as a covariate, and participant as a random effect. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 19 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 18 | 13 | 5
mg/dL | -52.23 [-61.54 to -42.93] | -57.43 [-64.21 to -50.64] | -18.22 [-44.69 to 8.25]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -34.01, 90% CI 2-sided [-56.14 to -11.88]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -39.20, 90% CI 2-sided [-61.15 to -17.26]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 5.20, 90% CI 2-sided [-4.28 to 14.67]

45. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 24 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Plasma glucose concentrations were obtained on Day -1 at pre meal (breakfast), 1, 3, 4 (pre lunch), 5, 7, 10 (pre dinner), 11, 13, 15 and 23 hours post breakfast meal and Day 24 at 1 (pre breakfast), 2, 4, 5 (pre lunch), 6, 8, 11 (pre dinner), 12, 14, 16, 24 hours post dose. The timing of samples on Day -1 are relative to the breakfast meal. Day 24 samples are relative to dosing. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with group, day and group by day interaction as fixed effects, baseline 24-hour WMG as a covariate, and participant as a random effect. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 24 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
mg/dL | -50.44 [-59.89 to -40.99] | -60.66 [-67.60 to -53.72] | -26.71 [-53.18 to -0.24]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -23.73, 90% CI 2-sided [-45.89 to -1.56]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -33.95, 90% CI 2-sided [-55.93 to -11.98]
Statistical Analysis 3: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 10.23, 90% CI 2-sided [0.56 to 19.89]

46. Secondary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Day 29 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: The 24-hour WMG was calculated as the area under the 24-hour glucose curve (AUC0-24hr) divided by 24 hours. Plasma glucose concentrations were obtained on Day -1 at pre meal (breakfast), 1, 3, 4 (pre lunch), 5, 7, 10 (pre dinner), 11, 13, 15 and 23 hours post breakfast meal and Day 29 at 1 (pre breakfast), 2, 4, 5 (pre lunch), 6, 8, 11 (pre dinner), 12, 14, 16, 24 hours post dose. The timing of samples on Day -1 are relative to the breakfast meal. Day 29 samples are relative to dosing. The change from baseline value for 24-hour WMG was calculated where baseline was the WMG before food and prior to treatment on Day 1. Individual change from baseline 24-hour WMG was analyzed in a linear mixed effects model with group, day and group by day interaction as fixed effects, baseline 24-hour WMG as a covariate, and participant as a random effect. WMG is presented as least squares mean with a 95% confidence interval.
Time Frame: Baseline (predose and before food on Day 1) and up to 24 hours post Day 29 dose
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM | Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM | Part 2: Placebo for MK-8521-T2DM
Number analyzed (Participants) | 16 | 11 | 5
mg/dL | -53.44 [-62.89 to -43.99] | -59.72 [-66.66 to -52.78] | -29.96 [-56.43 to -3.49]
Statistical Analysis 1: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -23.49, 90% CI 2-sided [-45.65 to -1.32]
Statistical Analysis 2: Comparison: Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM vs Part 2: Placebo for MK-8521-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = -29.76, 90% CI 2-sided [-51.74 to -7.79]
Statistical Analysis 3: Comparison: Part 2: MK-8521 64/120/180/240/300 µg/Day-T2DM vs Part 2: Liraglutide 0.6/1.2/1.8 mg/Day-T2DM; Test type: Other; Linear Mixed Effects Model; [statistical method as in outcome 37, analysis 1]; Difference of Least Squares Means = 6.27, 90% CI 2-sided [-3.39 to 15.93]

47. Secondary Outcome: Maximum Concentration (Cmax) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) and Non-Diabetic Overweight/Obese Participants in Part 2
Description: Cmax was the maximum observed concentration of MK-8521 in plasma after administration. Plasma samples were collected from predose to 120 hours postdose for determination of Cmax. Per protocol, Cmax in the non-diabetic overweight/obese participants was not measured on Days 19, 24, and 29 because they only received 14 days of treatment. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. Cmax is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 6, 10, 16, 24 hours post dose on Days 1, 7, 14, 19, 24 (T2DM) and Days 1 and 7 (Non-Diabetic Overweight/Obese); predose and 1, 2, 6, 10, 16, 24, 72, 96. and 120 hours post dose on Day 14 (Non-Diabetic Overweight/Obese) and Day 29 (T2DM).
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Part 2: MK-8521 64/120/180/240/300 μg/Day-T2DM: Type 2 diabetes mellitus (T2DM) participants received once daily subcutaneous MK-8521 titrated to 300 μg starting at 64 μg and increasing to 120 μg on Day 8, 180 μg on Day 15, 240 μg on Day 20, and 300 μg on Day 25. The total number of dosing days was 29.
- Part 2: MK-8521 64/120 μg/Day-Non-Diabetic Overweight/Obese: Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 titrated to 120 μg starting at 64 μg and increasing to 120 μg on Day 8. The total number of dosing days was 14.
Arm/Group | Part 2: MK-8521 64/120/180/240/300 μg/Day-T2DM | Part 2: MK-8521 64/120 μg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 8
nM
  Day 1 | 0.35 (48.0) | 0.411 (32.1)
  Day 7 | 0.719 (34.6) | 0.742 (38.7)
  Day 14 | 1.43 (35.8) | 1.72 (20.0)
  Day 19: number analyzed (Participants) | 18 | 0
  Day 19 | 2.27 (38.6) |
  Day 24: number analyzed (Participants) | 16 | 0
  Day 24 | 2.85 (33.1) |
  Day 29: number analyzed (Participants) | 16 | 0
  Day 29 | 3.14 (34.1) |

48. Secondary Outcome: Trough Concentration (Ctrough) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) and Non-Diabetic Overweight/Obese Participants in Part 2
Description: Ctrough was the lowest observed concentration of MK-8521 in plasma. Plasma samples were collected predose on Day 2 (sampled after the Day 1 dose and prior to Day 2 dose), 7, 14, 19, 24, and 29 for determination of Ctrough. Per protocol, Ctrough in the non-diabetic overweight/obese participants was not measured on Days 19, 24, and 29 because they only received 14 days of treatment. Individual values were natural log-transformed and evaluated with a linear-mixed effects model containing fixed effects for treatment, day, and treatment by day interaction, and a random effect for participant. Kenward and Roger's method was used to calculate the degree of freedom for the fixed effects. Ctrough is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose on Days 2 (sampled 24 hours after Day 1 dose) and 7, 14, 19, 24, and 29
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Arm/Group | Part 2: MK-8521 64/120/180/240/300 μg/Day-T2DM | Part 2: MK-8521 64/120 μg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 8
nM
  Day 1 | 0.331 (45.5) | 0.388 (32.8)
  Day 7 | 0.533 (32.7) | 0.492 (29.1)
  Day 14 | 1.07 (36.0) | 1.12 (21.8)
  Day 19: number analyzed (Participants) | 18 | 0
  Day 19 | 1.61 (33.8) |
  Day 24: number analyzed (Participants) | 16 | 0
  Day 24 | 2.02 (30.6) |
  Day 29: number analyzed (Participants) | 15 | 0
  Day 29 | 2.47 (29.9) |

49. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8521 for Type 2 Diabetes Mellitus (T2DM) and Non-Diabetic Overweight/Obese Participants in Part 2
Description: Tmax was the time required to reach the maximum concentration of MK-8521 in plasma. Plasma samples were collected from predose to 120 hours postdose for determination of Tmax. Per protocol, Tmax in the non-diabetic overweight/obese participants was not measured on Days 19, 24, and 29 because they only received 14 days of treatment. Tmax is presented as median with a full range.
Time Frame: as for outcome 47
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: MK-8521 64/120/180/240/300 μg/Day-T2DM | Part 2: MK-8521 64/120 μg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 18 | 8
Hours
  Day 1 | 16 [10 to 24] | 16 [10 to 24]
  Day 7 | 10 [1 to 16] | 10 [10 to 10]
  Day 14 | 6 [1 to 10] | 6 [6 to 10]
  Day 19: number analyzed (Participants) | 18 | 0
  Day 19 | 6 [6 to 10] |
  Day 24: number analyzed (Participants) | 16 | 0
  Day 24 | 6 [6 to 16] |
  Day 29: number analyzed (Participants) | 16 | 0
  Day 29 | 10 [1 to 24] |

50. Secondary Outcome: Apparent Terminal Half Life (t1/2) of MK-8521 on Day 29 for Type 2 Diabetes Mellitus (T2DM) Participants in Part 2
Description: t1/2 was the time required to divide the MK-8521 concentration by half after reaching pseudo-equilibrium. Plasma samples were collected from predose to 120 hours postdose for determination of t1/2. Per protocol, t1/2 was measured on Day 29 which is the longest time point for sampling for T2DM participants 1/2 is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 6, 10, 16, 24, 72, 96 and 120 hours post dose on Day 29
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: MK-8521 64/120/180/240/300 μg/Day-T2DM
Number analyzed (Participants) | 16
Hours | 15.4 (10.2)

51. Secondary Outcome: Apparent Terminal Half Life (t1/2) of MK-8521 on Day 14 for Non-Diabetic Overweight/Obese Participants in Part 2
Description: t1/2 was the time required to divide the MK-8521 concentration by half after reaching pseudo-equilibrium. Plasma samples were collected from predose to 24 hours postdose for determination of t1/2. Per protocol, t1/2 was measured on Day 14 which is the longest time point for sampling for non-diabetic overweight/obese participants 1/2 is presented as geometric mean and percent coefficient of variation of geometric mean.
Time Frame: Predose and 1, 2, 6, 10, 16, and 24 hours post dose on Day 14
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: MK-8521 64/120 μg/Day-Non-Diabetic Overweight/Obese
Number analyzed (Participants) | 8
Hours | 14.4 (10.8)

ADVERSE EVENTS:
Time Frame: Up to approximately 42 days for Part 1 and up to approximately 57 days for Part 2
Description: All participants that received ≥1 dose of study drug for adverse events (AEs) and all randomized participants for all-cause mortality. AEs and all-cause mortality are presented by individual dose received by participants during titration in an assigned study treatment sequence.
Groups:
- Part 2: MK-8521 64 μg/Day T2DM: Type 2 Diabetes Mellitus (T2DM) participants received once daily subcutaneous MK-8521 64 µg on Days 1 to 7 as part of the MK-8521 64/120/180/240/300 µg treatment sequence.
- Part 2: MK-8521 120 μg/Day T2DM: T2DM participants received once daily subcutaneous MK-8521 120 µg on Days 8 to 14 as part of the MK-8521 64/120/180/240/300 µg treatment sequence.
- Part 2: MK-8521 180 μg/Day T2DM: T2DM participants received once daily subcutaneous MK-8521 180 µg on Days 15 to 19 as part of the MK-8521 64/120/180/240/300 µg treatment sequence.
- Part 2: MK-8521 240 μg/Day T2DM: T2DM participants received once daily subcutaneous MK-8521 240 µg on Days 20 to 24 as part of the MK-8521 64/120/180/240/300 µg treatment sequence.
- Part 2: MK-8521 300 μg/Day T2DM: T2DM participants received once daily subcutaneous MK-8521 300 µg on Days 25 to 29 as part of the MK-8521 64/120/180/240/300 µg treatment sequence.
- Part 2: Liraglutide 0.6 mg/Day T2DM: T2DM participants received once daily subcutaneous liraglutide 0.6 mg on Days 1 to 7 as part of the liraglutide 0.6/1.2/1.8 mg treatment sequence.
- Part 2: Liraglutide 1.2 mg/Day T2DM: T2DM participants received once daily subcutaneous liraglutide 1.2 mg on Days 8 to 14 as part of the liraglutide 0.6/1.2/1.8 mg treatment sequence.
- Part 2: Liraglutide 1.8 mg/Day T2DM: T2DM participants received once daily subcutaneous liraglutide 1.8 mg on Days 15 to 29 as part of the liraglutide 0.6/1.2/1.8 mg treatment sequence.
- Part 2: MK-8521 64 μg/Day-Non-Diabetic Overweight/Obese: Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 64 µg on Days 1 to 7 as part of the MK-8521 64/120 µg treatment sequence.
- Part 2: MK-8521 120 μg/Day-Non-Diabetic Overweight/Obese: Non-diabetic overweight/obese participants received once daily subcutaneous MK-8521 120 µg on Days 8 to 14 as part of the MK-8521 64/120 µg treatment sequence.
Arm/Group | Part 1: MK-8521 64 μg/Day | Part 1: MK-8521 120 μg/Day | Part 1: MK-8521 34 μg/Day | Part 1: MK-8521 72 μg/Day | Part 1: Liraglutide 0.6 mg/Day | Part 1: Liraglutide 1.2 mg/Day | Part 1: Liraglutide 1.8 mg/Day | Part 1: Placebo for MK-8521 | Part 2: MK-8521 64 μg/Day T2DM | Part 2: MK-8521 120 μg/Day T2DM | Part 2: MK-8521 180 μg/Day T2DM | Part 2: MK-8521 240 μg/Day T2DM | Part 2: MK-8521 300 μg/Day T2DM | Part 2: Liraglutide 0.6 mg/Day T2DM | Part 2: Liraglutide 1.2 mg/Day T2DM | Part 2: Liraglutide 1.8 mg/Day T2DM | Part 2: Placebo for MK-8521-T2DM | Part 2: MK-8521 64 μg/Day-Non-Diabetic Overweight/Obese | Part 2: MK-8521 120 μg/Day-Non-Diabetic Overweight/Obese
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/7 | 0/8 | 0/8 | 0/11 | 0/11 | 0/8 | 0/8 | 0/18 | 0/18 | 0/18 | 0/18 | 0/15 | 0/14 | 0/13 | 0/13 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/7 | 0/8 | 0/8 | 0/11 | 0/11 | 0/8 | 0/8 | 0/18 | 0/18 | 0/18 | 1/18 | 0/15 | 0/14 | 0/13 | 0/13 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/9 | 5/7 | 1/8 | 4/8 | 2/11 | 7/11 | 2/8 | 5/8 | 8/18 | 14/18 | 6/18 | 13/18 | 8/15 | 8/14 | 8/13 | 12/13 | 3/6 | 2/8 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-8521 64 μg/Day (N=9) | Part 1: MK-8521 120 μg/Day (N=7) | Part 1: MK-8521 34 μg/Day (N=8) | Part 1: MK-8521 72 μg/Day (N=8) | Part 1: Liraglutide 0.6 mg/Day (N=11) | Part 1: Liraglutide 1.2 mg/Day (N=11) | Part 1: Liraglutide 1.8 mg/Day (N=8) | Part 1: Placebo for MK-8521 (N=8) | Part 2: MK-8521 64 μg/Day T2DM (N=18) | Part 2: MK-8521 120 μg/Day T2DM (N=18) | Part 2: MK-8521 180 μg/Day T2DM (N=18) | Part 2: MK-8521 240 μg/Day T2DM (N=18) | Part 2: MK-8521 300 μg/Day T2DM (N=15) | Part 2: Liraglutide 0.6 mg/Day T2DM (N=14) | Part 2: Liraglutide 1.2 mg/Day T2DM (N=13) | Part 2: Liraglutide 1.8 mg/Day T2DM (N=13) | Part 2: Placebo for MK-8521-T2DM (N=6) | Part 2: MK-8521 64 μg/Day-Non-Diabetic Overweight/Obese (N=8) | Part 2: MK-8521 120 μg/Day-Non-Diabetic Overweight/Obese (N=8)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-8521 64 μg/Day (N=9) | Part 1: MK-8521 120 μg/Day (N=7) | Part 1: MK-8521 34 μg/Day (N=8) | Part 1: MK-8521 72 μg/Day (N=8) | Part 1: Liraglutide 0.6 mg/Day (N=11) | Part 1: Liraglutide 1.2 mg/Day (N=11) | Part 1: Liraglutide 1.8 mg/Day (N=8) | Part 1: Placebo for MK-8521 (N=8) | Part 2: MK-8521 64 μg/Day T2DM (N=18) | Part 2: MK-8521 120 μg/Day T2DM (N=18) | Part 2: MK-8521 180 μg/Day T2DM (N=18) | Part 2: MK-8521 240 μg/Day T2DM (N=18) | Part 2: MK-8521 300 μg/Day T2DM (N=15) | Part 2: Liraglutide 0.6 mg/Day T2DM (N=14) | Part 2: Liraglutide 1.2 mg/Day T2DM (N=13) | Part 2: Liraglutide 1.8 mg/Day T2DM (N=13) | Part 2: Placebo for MK-8521-T2DM (N=6) | Part 2: MK-8521 64 μg/Day-Non-Diabetic Overweight/Obese (N=8) | Part 2: MK-8521 120 μg/Day-Non-Diabetic Overweight/Obese (N=8)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Change of bowel habit (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (6) | 6 (6) | 0 (0) | 1 (1) | 3 (3) | 5 (6) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 2 (4) | 4 (4) | 0 (0) | 5 (6) | 1 (1) | 5 (7) | 2 (3) | 5 (6) | 1 (1) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application site irritation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site injury (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site macule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wrinkling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.